CLINICAL TRIAL: NCT01433185
Title: Improving Uptake of Early Infant Diagnosis of HIV for PMTCT: a Randomized Trial of a Text Messaging Intervention
Brief Title: Improving Uptake of Early Infant Diagnosis of HIV for the Prevention of Mother-to-child Transmission of HIV
Acronym: SMS4PMTCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Kenya Medical Research Institute (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Thomas Odeny, Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 41186-E/G
Record Dates: First submitted 2011-09-12; First posted 2011-09-13 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: HIV Infections; Acquired Immunodeficiency Syndrome
Keywords: PMTCT; SMS; HIV Infections; Acquired Immunodeficiency Syndrome; Prevention & Control; Patient Compliance; Cellular Phone; Randomized Controlled Trial
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Patient Compliance | interventions — Spermine Synthase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Text message (SMS) (Experimental): Text messages sent to women before and after delivery
  Interventions: Other: Text message
- Usual care (current standard of care) (No Intervention): Current standard of care for women enrolled in PMTCT programs

INTERVENTIONS:
Other: Text message — Text messages sent to women before and after delivery
  Other Names: SMS, short message service, text messaging
  Arms: Text message (SMS)

SUMMARY:
Early accurate diagnosis is one of the first crucial steps in care for infants born to HIV-infected mothers. Early initiation of antiretroviral therapy (ART) relies upon early diagnosis and results in significant reductions in infant morbidity and mortality. There is little information on evidence-based interventions that specifically target improved attendance of postpartum clinic visits and subsequent infant HIV testing in the context of prevention of mother-to-child transmission of HIV (PMTCT) programs. The investigators propose a randomized controlled trial to examine the effect of text messages sent to women enrolled in PMTCT programs on adherence to postpartum clinic visits and uptake of early infant diagnosis by DNA polymerase chain reaction (PCR). This study seeks to test the hypotheses that (a) text messages sent to women enrolled in PMTCT will improve their attendance at the postnatal clinic within the first 6-8 weeks after childbirth; and (b) text messages sent to women enrolled in PMTCT programs will increase uptake of DNA PCR HIV testing at 6-8 weeks among infants exposed to HIV. This study will evaluate a novel strategy to improve adherence to postnatal clinic visits and increase the uptake of infant HIV testing. If proven superior to standard care, the proposed intervention can be easily scaled-up and integrated into existing healthcare systems in resource-limited settings. Findings from this study will provide randomized trial evidence to inform HIV prevention program planners and implementers. This study will also provide further information on the feasibility of using mobile phone-based technology for public health interventions in resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

* age at least 18 years
* report ability to read SMS
* ≥ 28 weeks gestation or delivery at study clinic on day of enrollment
* HIV positive women enrolled in the PMTCT program
* have access to a mobile phone (personal or partner's if HIV serostatus disclosed to partner)
* willing to receive SMS messages from the study
* planning to remain in the study area (Nyanza province) for the duration of the study

Exclusion Criteria:

* age less than 18 years old
* women who share phones with partners but HIV status not disclosed to partners
* intention to deliver at a non-study hospital

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2012-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Proportion of women who attend postnatal clinic within 6-8 weeks postpartum | 6-8 weeks after delivery
Proportion of infants tested for HIV by DNA PCR | 6-8 weeks after delivery

SECONDARY OUTCOMES:
Infant adherence to antiretroviral prophylaxis | Up to 6 weeks after delivery
Time to post-natal clinic return | Up to 8 weeks after delivery
Maternal adherence to antiretroviral prophylaxis | Up to 8 weeks after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Odeny, MBChB, MPH, Principal Investigator — University of Washington/Kenya Medical Research Institute; R Scott McClelland, MD, MPH, Study Chair — University of Washington; Craig R Cohen, MD, MPH, Study Chair — University of California, San Francisco; Carol Camlin, PhD, Study Chair — University of California, San Francisco; Elizabeth A Bukusi, MBChB, MMed, MPH, PhD, Study Chair — Kenya Medical Research Institute
Locations (1):
- Kenya Medical Research Institute, Family AIDS Care and Education Services, Kisumu, Nyanza, Kenya

REFERENCES:
- [Result] Odeny TA, Bukusi EA, Cohen CR, Yuhas K, Camlin CS, McClelland RS. Texting improves testing: a randomized trial of two-way SMS to increase postpartum prevention of mother-to-child transmission retention and infant HIV testing. AIDS. 2014 Sep 24;28(15):2307-12. doi: 10.1097/QAD.0000000000000409. PMID 25313586
- [Result] Odeny TA, Newman M, Bukusi EA, McClelland RS, Cohen CR, Camlin CS. Developing content for a mHealth intervention to promote postpartum retention in prevention of mother-to-child HIV transmission programs and early infant diagnosis of HIV: a qualitative study. PLoS One. 2014 Sep 2;9(9):e106383. doi: 10.1371/journal.pone.0106383. eCollection 2014. PMID 25181408